CLINICAL TRIAL: NCT05766332
Title: Developing Novel Tools for Determining Risk of Respiratory Complications Following Hematopoietic Stem Cell Transplant
Brief Title: Evaluating Clinical Evaluation Tools for Predicting Risk of Complications After Hematopoietic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-000913; NCI-2022-01589 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-000913 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2023-02-22; First posted 2023-03-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (clinical evaluation, record review): Patients undergo a clinical evaluation consisting of a six-minute walk test, hand grip strength test, and gait speed test on study. Patients' medical records are also reviewed for a year on study.
  Interventions: Other: Clinical Evaluation; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Clinical Evaluation — Undergo clinical evaluation
  Other Names: Clinical Assessment
Other: Electronic Health Record Review — Medical records reviewed

SUMMARY:
This study evaluates whether clinical evaluation tools such as the six-minute walk test, hand grip strength test, and gait speed test, are useful in predicting risk of complications in patients undergoing hematopoietic stem cell transplants (HCT). Being able to predict who is at increased risk of post-HCT complications can help better inform patients and providers on the risks and benefits of undergoing HCT and determine whether certain patients should have closer post-HCT monitoring due to an increased risk of complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop novel pre-transplant tools for determining risk of post-HCT pulmonary complications.

OUTLINE: This is an observational study.

Patients undergo a clinical evaluation consisting of a six-minute walk test, hand grip strength test, and gait speed test on study. Patients' medical records are also reviewed for a year on study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >= 18 years old)
* Undergoing evaluation for autologous or allogeneic bone marrow transplant (HCT) at Mayo Clinic Rochester
* Scheduled for pre-HCT pulmonary function test by the primary team

Exclusion Criteria:

* Limited mobility requiring use of gait aid or wheelchair
* Fall risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing evaluation for autologous or allogeneic bone marrow transplant.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Pulmonary complication following hematopoietic stem cell transplant (HCT) | Up to 1 year after transplant
  Pulmonary complications may include but are not limited to: infection, HCT-specific lung injury syndromes, acute respiratory distress syndrome, pulmonary graft versus host disease. Univariable analysis will be first used to identify potential factors that predict post-HCT pulmonary complications. All possible factors will then be included in multivariable analysis. Will also specifically test whether the six-minute walk test, grip strength and gait speed add additional significance to pulmonary complications and the statistic model after including pulmonary function test results.

SECONDARY OUTCOMES:
100-day mortality | At 100 days after transplant
  Analyses similar to those for the primary outcome will be conducted.
1 year mortality | At 1 year after transplant
  Analyses similar to those for the primary outcome will be conducted.
Relapse-free survival | At 1 year after transplant
  Analyses similar to those for the primary outcome will be conducted.
Hospital or intensive care unit admission post-HCT | Up to 1 year after transplant
  Will specifically test whether the six-minute walk test, grip strength and gait speed add additional significance to pulmonary complications and the statistic model after including pulmonary function test results.
Need for noninvasive or invasive mechanical ventilation | Up to 1 year after transplant
  Will specifically test whether the six-minute walk test, grip strength and gait speed add additional significance to pulmonary complications and the statistic model after including pulmonary function test results.

CONTACTS AND LOCATIONS:
Overall Officials: Hemang Yadav, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials